CLINICAL TRIAL: NCT00180583
Title: Vision II: Non Randomized French Evaluation of GALILEO Intravascular Radiotherapy System in Patients With de Novo Coronary Arteries Lesions by Restenosis on Angioplasty or Restenosis on Endoprosthesis
Brief Title: Vision II: Evaluation of GALILEO Intravascular Radiotherapy System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Matt Kiely, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vision II v. 1.1 07/02/2002
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (1):
- 1 (Experimental): Treatment of single or multivessel long diffuse coronary stenosis with the Guidant GALILEO Intravascular Radiotherapy System
  Interventions: Device: Guidant GALILEO Intravascular Radiotherapy System

INTERVENTIONS:
Device: Guidant GALILEO Intravascular Radiotherapy System — Treatment of single or multivessel long diffuse coronary stenosis with the Guidant GALILEO Intravascular Radiotherapy System

SUMMARY:
To assess the safety and effectiveness of intravascular brachytherapy for the treatment of intrastent restenosis of coronary lesions with the Galileo system

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the cardiac events (MACE) and adverse extra cardiac events at 6 month follow up and up to 24 months for the patients treated with Galileo system

ELIGIBILITY:
Inclusion Criteria:

* Patient with angor, patients with only one de novo lesion. Target zone must be < 52 mm, artery section must be < 3,7mm and > 2,25 mm

Exclusion Criteria:

* Vessel with extremely tortuous proximal segment, lesion with angulous segments (>90°) Unstable ventricular arrhythmia, dialysis, MI within the last 72 hours etc…

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2002-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
MACE | 6 months

SECONDARY OUTCOMES:
All adverse cardiac or extra cardiac events | 24-month

CONTACTS AND LOCATIONS:
Overall Officials: Jacques BERLAND, MD, Principal Investigator — Clinique St Hilaire, Rouen, France
Locations (1):
- Clinique St. Hilaire, Rouen, France